CLINICAL TRIAL: NCT03212651
Title: A Phase II Study Evaluating Neoadjuvant Pembrolizumab Monotherapy in Patients With Muscle-Invasive Bladder Cancer to Explore in Vivo the Mechanisms of Action of Pembrolizumab
Brief Title: Study Evaluating Neoadjuvant Pembrolizumab Monotherapy in Patients With Muscle-Invasive Bladder Cancer to Explore in Vivo the Mechanisms of Action of Pembrolizumab
Acronym: PANDORE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-002537-29; 2016/2432 (Other: CSET number)
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with MIBC (Muscle Invasive Bladder Cancer) (Experimental): Cisplatinum-ineligible patients with muscle-invasive bladder cancer
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200mg IV infusion

SUMMARY:
monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2; Recent phase I trial provided evidence of activity of pembrolizumab in advanced platinum-resistant metastatic urothelial carcinoma; Recent phase 3 trial showed an overall survival benefit in patients treated with pembrolizumab in a trial comparing pembrolizumab to chemotherapy in patients who failed first-line platinum-based chemotherapy Neoadjuvant chemotherapy followed by radical cystectomy is the standard of care for cisplatinum-eligible non-metastatic MIBC patients; Many patients with MIBC are unfit for cisplatin-based combination treatment; Given its safety profile, pembrolizumab may be used in unfit patients; Neo-adjuvant setting is a unique opportunity to assess mechanisms of action of pembrolizumab in human

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial.
2. Be >/= 18 years of age on day of signing informed consent.
3. Histologically confirmed muscle invasive transitional cell carcinoma of the bladder (Note: urothelial carcinoma invading into the prostatic stroma with no histologic muscle invasion is allowed, provided that the extent of disease is confirmed via imaging and/or EUA. Patients with mixed histologies are required to have a dominant transitional cell pattern)
4. Clinical stage T2-T4a N0/X M0 disease according to TNM classification (within 4 weeks before registration)
5. Medically appropriate candidate for radical cystectomy as per urologic oncologist
6. Representative formalin-fixed paraffin embedded (FFPE) bladder tumor samples with an associated pathology report that are determined to be available and sufficient for central testing. If an insufficient amount of tumor tissue is available prior to the start of the screening phase, subjects must consent to allow the acquisition of additional tumor tissue for performance of central testing.
7. Patients who refuse neoadjuvant cisplatin based chemotherapy or in whom neoadjuvant cisplatin based therapy is not appropriate for the following conditions:

   1. ECOG performance status of 2
   2. Creatinine clearance (calculated according to MDRD formula or measured) less than 1mL/s
   3. CTCAE version 4.0, grade 2 or above audiometric hearing loss
   4. CTCAE version 4.0, grade 2 or above peripheral neuropathy
8. Adequate bone marrow function obtained within 14 days before registration

   1. Absolute neutrophil count ≥ 1,500/mm3
   2. Hb ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)
   3. Platelet count ≥ 100,000/mm3
9. Adequate organ function obtained within 14 days before registration

   1. Bilirubin ≤ 1.5 times upper limit of normal (ULN) or Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
   2. Alkaline phosphatase ≤ 2 x upper limit of normal (ULN);
   3. AST and ALT ≤2.5 x upper limit of normal (ULN);
   4. Creatinine clearance > 30 ml/min according to MDRD formula
   5. Albumin >2.5 mg/dL
10. Adequate Coagulation function

    1. International Normalized ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
    2. Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
11. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 14 days prior to the first dose of study treatment. Both sexually active females and males (and their female partners) patients must agree to use two methods of highly effective contraception, one of them being a barrier method, or to abstain from sexual activity during the study and for at least 4 months after last study drug administration.
12. Patient affiliated to a social security regimen or beneficiary of the same

Exclusion Criteria:

1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks before the first dose of study treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of systemic immunosuppressive therapy within 7 days prior to the first dose of study treatment (except local/topical or aerosol steroids)
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients
5. Has had a prior monoclonal antibody within 4 weeks or 5 halflife time (whatever the shortest) prior to the first dose of study treatment or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior intra-venous chemotherapy, targeted small molecule therapy, or radiation therapy for bladder cancer
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
8. Has an active autoimmune / immune mediated inflammatory disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
9. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
10. Has an active infection requiring systemic therapy.
11. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
12. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
13. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
14. Positive for Human Immunodeficiency Virus (HIV) antibody testing
15. Active or chronic hepatitis C and/or B infection. Patients with past/resolved HBV infection (defined as the presence of antihepatitis B core antibody, IgG anti-HBs +) are eligible. HBV DNA should be obtained in these patients prior to the first dose of study treatment. Patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA
16. Has received a live attenuated vaccine within 30 days prior to the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Pathologic complete response rate | Up to 1 month
  defined as the absence of carcinoma (pT0 disease) and the absence of microscopic lymph node metastases (N0) on the final cystectomy specimen in PD-L1 positive patients and PD-L1 negative patients

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: Undecided